CLINICAL TRIAL: NCT03494296
Title: A Prospective Study of Low-dose Decitabine Combined With COP Regimen in the Treatment of Relapsed and Refractory DLBCL
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Principal Investigator, Shuye Wang, Director of the lymphoma ward, First Affiliated Hospital of Harbin Medical University
Other Study IDs: Organization:FirstAHHarbinMU
Record Dates: First submitted 2018-03-19; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open, multi-center, prospective: All enrolled and relapsed patients received D-COP regimen chemotherapy
  Interventions: Drug: patients received D-COP regimen chemotherapy

INTERVENTIONS:
Drug: patients received D-COP regimen chemotherapy — patients received D-COP regimen chemotherapy

SUMMARY:
Decitabine is a cytosine analogue and is a specific DNA methyltransferase (DNMT) inhibitor. It directly inhibits DNMT by phosphorylating DNA and inhibits DNMT, thereby reversing DNA methylation and inducing tumor cells to Normal cell differentiation or induction of tumor cell apoptosis.Diffuse large B-cell lymphoma (DLBCL) is the most common pathological type in non-Hodgkin's lymphoma. The first-line chemotherapy regimen using Rituximab+Cyclophosphamide+Doxorubicin +Vincristine+Bonisone（R-CHOP）significantly increases the remission rate and disease-free survival of patients with DLBCL, but it is difficult to partially relapse. Long-term remission and survival rates in treating patients are not satisfactory.Due to the greater cardiac toxicity of adriamycin, more patients can not be uncomfortable, so the COP program is also widely used in patients with DLBCL, and achieved a good response rate.In 2008, the FDA had approved decitabine for the demethylation treatment of Myelodysplastic syndrome（MDS）. Over the years, good initial remission rates and better long-term survival rates have been achieved in patients with MDS.There are also a variety of clinical trials of decitabine for patients with solid tumors that have achieved significant clinical efficacy.Due to the high side effects of high-dose decitabine, patient tolerance is poor. Therefore, the purpose of this study was to evaluate the efficacy and safety of low-dose decitabine combined with Cyclophosphamide+Vindesine+Bonisone(COP) regimen (D-COP) 4-6 course of treatment for relapsed and refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Decitabine is a cytosine analogue and is a specific DNA methyltransferase (DNMT) inhibitor. It directly inhibits DNMT by phosphorylating DNA and inhibits DNMT, thereby reversing DNA methylation and inducing tumor cells to Normal cell differentiation or induction of tumor cell apoptosis. High concentrations of decitabine inhibit DNA synthesis, exert its cytotoxic effects, and induce cell death; low concentrations of decitabine inactivate DNMT and demethylate some hypermethylated CpG islands in tumor suppressor genes. To activate the silencing tumor suppressor gene and exert its effect of inhibiting tumor growth to achieve anti-tumor effects.

Epigenetics plays an important role in the occurrence and development of tumors and is a hot topic in recent years. Methylation of DNA is the main form of epigenetic information. Normal methylation plays an important role in maintaining the normal functions of cells and organs and in the development, differentiation, growth, and aging of the body. However, the abnormal participation of cell epigenetics can directly affect the overexpression of tumor cells, which leads to the occurrence and development of tumor cells.

Diffuse large B-cell lymphoma (DLBCL) is the most common pathological type in non-Hodgkin's lymphoma. The first-line chemotherapy regimen using R-CHOP significantly increases the remission rate and disease-free survival of patients with DLBCL, but it is difficult to partially relapse. Long-term remission and survival rates in treating patients are not satisfactory.Due to the greater cardiac toxicity of adriamycin, more patients can not be uncomfortable, so the COP program is also widely used in patients with DLBCL, and achieved a good response rate.In 2008, the FDA had approved decitabine for the demethylation treatment of MDS. Over the years, good initial remission rates and better long-term survival rates have been achieved in patients with MDS.There are also a variety of clinical trials of decitabine for patients with solid tumors that have achieved significant clinical efficacy.Due to the high side effects of high-dose decitabine, patient tolerance is poor. Therefore, the purpose of this study was to evaluate the efficacy and safety of low-dose decitabine combined with COP regimen (D-COP) 4-6 course of treatment for relapsed and refractory diffuse large B-cell lymphoma.

In summary, this study will select relapsed refractory high-risk patients, previous studies have confirmed that the COP program can make a good effect in most patients, also confirmed the demethylation of decitabine in other tumors Therefore, whether the treatment of low-dose decitabine combined with COP regimen for DLBCL can improve the prognosis is worth looking forward to. At present, there are few researches on the treatment of DLBCL with low-dose decitabine at home and abroad. The purpose of this study is to explore whether low-dose decitabine combined with COP regimen as a treatment for patients with relapsed and refractory DLBCL can improve the relapse-refractory DLBCL. The patient's prognosis, and hope to explore through a stratified analysis which group of patients benefit more from it.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology confirmed as DLBCL.
2. Relapsed and refractory patients.
3. Age ≥ 18 years old.
4. ECOG ≥ 3.
5. Women are not lactating, not pregnant, and agree not to become pregnant during the study period and within the next 12 months. Male patients agree that their spouse is not pregnant during the study period and within the next 12 months。
6. There is an assessable lesion (lymph node diameter ≥ 1.0cm; or a dermatologic lesion that can be assessed by a physical examination)Signed informed consent

Exclusion Criteria:

1. Bone marrow involvement and lymphoma cells ≥ 25%.
2. Severe abnormal liver and kidney function (alanine aminotransferase, bilirubin, creatinine> 3 times the upper limit of normal).
3. Uncontrolled active infections.
4. Organic heart disease and clinical symptoms or abnormal heart function (NYHA ≥ 2).
5. Simultaneous presence of other tumors.
6. Other psychological conditions that prevent patients from participating in the study or signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Plans to enroll 150 cases within 2 years
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A Prospective Study of Low-dose Decitabine Combined With COP Regimen in the Treatment of Relapsed and Refractory DLBCL | From March 1, 2018 to December 31, 2020
  Primary end point:
  Using 5-year progression-free survival (PFS) as an index to evaluate the clinical effect of low-dose decitabine combined with COP chemotherapy.clinical efficacy of low-dose decitabine combined with COP regimen chemotherapy.
  Efficacy assessment criteria:2007 revised standards for international lymphoma efficacy: J Clin Oncol 2007;25(5):579-586.

CONTACTS AND LOCATIONS:
Overall Officials: Shuye Wang, PhD, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Department of Hematology, Lymphoma Ward, Harbin, Heilongjiang, China